CLINICAL TRIAL: NCT03462199
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Parallel Study to Evaluate the Efficacy of the Investigational Products on Complete Spontaneous Bowel Movements in Participants Who Normally Have ≤ 3 Complete Spontaneous Bowel Movements Per Week But Are Otherwise Healthy
Brief Title: Evaluating Efficacy of Investigational Products on Spontaneous Bowel Movements in Healthy People With ≤ 3 Complete Weekly Spontaneous Bowel Movements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AIDP, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18ACHA
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2019-07

CONDITIONS: Functional Constipation; Healthy
Keywords: Kiwi; Constipation; Bowel Movements; Healthy; Functional Constipation
MeSH Terms: conditions — Constipation | interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo controlled, parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo (microcrystalline cellulose)
- Actazin High Dose (Experimental)
  Interventions: Dietary Supplement: Actazin (green kiwi powder) High Dose
- Actazin Low Dose (Experimental)
  Interventions: Dietary Supplement: Actazin (green kiwi powder) Low Dose
- Control Formula (Active Comparator)
  Interventions: Dietary Supplement: Control Formula (Actazin green kiwi powder + PreticX prebiotic)
- Livaux High Dose (Experimental)
  Interventions: Dietary Supplement: Livaux (gold kiwi powder) High Dose
- Livaux Low Dose (Experimental)
  Interventions: Dietary Supplement: Livaux (gold kiwi powder) Low Dose

INTERVENTIONS:
Dietary Supplement: Actazin (green kiwi powder) High Dose — Participants will consume 4 capsules (600 mg green kiwi powder) daily for 28-days
  Arms: Actazin High Dose
Dietary Supplement: Actazin (green kiwi powder) Low Dose — Participants will consume 4 capsules (150 mg green kiwi powder) daily for 28-days
  Arms: Actazin Low Dose
Dietary Supplement: Control Formula (Actazin green kiwi powder + PreticX prebiotic) — Participants will consume 4 capsules (150 mg green kiwi powder + 250 mg PreticX prebiotic) daily for 28-days
  Arms: Control Formula
Dietary Supplement: Livaux (gold kiwi powder) High Dose — Participants will consume 4 capsules (600 mg gold kiwi powder) daily for 28-days
  Arms: Livaux High Dose
Dietary Supplement: Livaux (gold kiwi powder) Low Dose — Participants will consume 4 capsules (150 mg gold kiwi powder) daily for 28-days
  Arms: Livaux Low Dose
Dietary Supplement: Placebo (microcrystalline cellulose) — Participants will consume 4 capsules containing no active ingredients daily for 28-days
  Arms: Placebo

SUMMARY:
Low and High doses of Actazin and Livaux will be compared against a control formula and placebo to evaluate how each investigational study product effects complete spontaneous bowel movements in healthy adults that currently experience less than or equal to 3 complete spontaneous bowel movements per week. During the 28-day study period, it is hypothesized that participants consuming Acatzin, Livaux, or control formula will have an increased number of complete spontaneous bowel movements when compared to participants consuming the placebo. It is hypothesized that participants consuming Actazin or Livaux will respond more than participants consuming the control formula. It is hypothesized that participants consuming Actazin or Livaux will have a favorable microbiome change than placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 60 years of age, inclusive at baseline
* Female participant is not of child bearing potential, defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) or,

Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. All birth control must have been in use for a minimum of three months and the participant must have one regular menstrual cycle in the last 30 days. Acceptable methods of birth control include:

* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method
* Intrauterine devices
* Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
* Vasectomy of partner (shown successful as per appropriate follow-up)
* Body mass index (BMI) between 19 and 29.9 ±1 kg/m2 at screening, inclusive
* Participants must have the following criteria based on participant self-reporting:
* Self-reported ≤ 3 CSBMs per week at screening and confirmed in the BHD during the run-in period for enrolment at baseline
* People who are not regular consumers of, high fibre diets, yoghurt, fermented foods such as kimchi, kombucha, sauerkraut etc.
* Fasting blood glucose ≤6.0 mmol/L at screening
* Agree to refrain from the consumption high-fiber dietary supplements including Metamucil, Benefibre, and Phloe
* Agree to refrain from the consumption of fresh kiwifruit 2-weeks prior to and during the study
* Agree to maintain their habitual food and beverage intakes
* Agree to maintain current physical activity patterns
* Agree to avoid overseas travel for the duration of the study due to the impact this may have on diet and gastrointestinal health
* Healthy as determined by laboratory results, medical history, and physical exam as assessed by the Qualified Investigator
* Willingness to complete questionnaires, records, and diaries associated with the study, collect stool samples, and to complete all clinic visits
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breast feeding, or planning to become pregnant during the trial
* Participation in a clinical research trial within 30 days prior to randomization
* Blood donation during the study or within 30 days of completing the study
* Vegan, raw food, or very high-fiber diet, including regular consumption of foods labeled as supplemented with fiber.
* Weight loss of >5% within the past 3 months
* Frequent use of laxatives defined as greater than once per week.
* Use of medications such as antibiotics that have major impact on gut microbes 2 months prior to baseline and as assessed case by case by the QI
* Use of probiotic and prebiotic dietary supplements.
* Regular intake of nonsteroidal anti-inflammatory drugs (NSAIDs), steroids, or other anti-inflammatory medications
* Use of medications for constipation and or Diarrhea as assessed by QI
* Allergy or sensitivity to kiwifruit or other test product ingredients
* Prior surgery for weight loss (lap band or gastric bypass)
* Gastrointestinal alarm symptoms including blood in stools, frequent diarrhea, and unremitting abdominal pain, and major diseases of the gastrointestinal tract (such as IBS, Crohn's, etc.), pulmonary or endocrine systems, or other GI abnormalities
* Gastroparesis or lactose intolerance
* Current, or history of, thyroid disease
* Uncontrolled hypertension (SBP ≥160 mmHg) assessed by QI
* Renal, hepatic, pancreatic, or biliary impairment or disease as disclosed or detected (if applicable) by chemistry and hematology taken at screening
* Current, or history of, bleeding/blood disorders
* Type I and Type II diabetes
* Autoimmune disease or immuno-compromised (i.e. HIV positive, use of anti-rejection medication, rheumatoid arthritis, Hepatitis B/C positive)
* Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis will be considered as per the QI's opinion
* Clinically significant abnormal laboratory results at screening
* Alcohol or drug abuse within the last 6 months
* Participants with a history of cigarette smoking within the past 5 years.
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the qualified investigator's opinion may adversely affect the participant's ability to complete the study or its measures or which may pose significant risk to the participant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
The change in complete spontaneous bowel movements between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and Placebo | 28 days
  Assessed by the daily bowel habits diary. A complete spontaneous bowel movements is defined as bowel movements that are both complete and spontaneous.

SECONDARY OUTCOMES:
The change in spontaneous bowel movements per week between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed using the daily bowel habits diary
The change in stool form between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed by the Brstiol Stool Scale (BSS). BSS scores are a measure of stool form. It is on a scale of 1-7, 1 = highly constipated; 7 = diarrhea. A score of type 3-4 are considered normal and movement towards these scores are indicative of healthier bowel functions.
The change in interval between bowel movements in hours between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed using the daily bowel habits diary
The change in blood calcium levels between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed by fasting blood sample analysis
The change in fasting glucose levels between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed by fasting blood sample analysis
The change in the Patient Assessment of Constipation Symptoms Questionnaire (PAC-SYM) between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed by the participants answers to the PAC-SYM questions which assess the severity of patient-reported symptoms of constipation. It is ona scale of 0-4 ( 0= symptoms absent and 4 = severe symptoms.
The change in the Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QoL) between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed by the participants answers to the PAC-QoL questions. Effect on quality of life is measured on a scale of 0 - 4 (0= no effect on quality of life, and 4 = negative effect on quality of life
The change in gut microbiome between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed by fecal sample analysis
The percentage of early and late responders to Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed by the bowel habits diary
The difference in the Bowel Regularity Index Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo. | 28 days
  Assessed by the Bowel Regularity Index questionnaire in which participants were provided with a series of twelve statements and asked to score each. Scoring for this index is based on a five-point scale for each question, from strongly disagree (0) to strongly agree (5).

OTHER OUTCOMES:
Adverse events (AEs) | up to 45 days for non-supplement emergent AE's, and 28-days for supplement emergent AE's
  The incidence of adverse events (AEs) between Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo.
Systolic and diastolic blood pressure. | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on systolic and diastolic blood pressure.
Heart rate. | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on heart rate.
Body weight. | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on body weight.
Body mass index (BMI). | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on body mass index (BMI).
Fasting glucose | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on fasting glucose
Alanine Transaminase | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Alanine Transaminase
Aspartate Transaminase | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Aspartate Transaminase
Total Bilirubin | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Total Bilirubin
Creatinine | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Creatinine
Sodium ion | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Sodium ion
Potassium ion | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Potassium ion
Chloride ion | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Chloride ion
Estimated Glomerular Filtration Rate (eGFR) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Estimated Glomerular Filtration Rate (eGFR)
White Blood Cell Count | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on White Blood Cell Count
Red Blood Cell | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Red Blood Cell
Hemoglobin | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Hemoglobin
Hematocrit | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Hematocrit
Platelet Count | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Platelet Count
Mean corpuscular Volume (MCV) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Mean corpuscular Volume (MCV)
Mean corpuscular Hemoglobin (MCH) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Mean corpuscular Hemoglobin (MCH)
Mean corpuscular Hemoglobin Concentration (MCHC) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Mean corpuscular Hemoglobin Concentration (MCHC)
Absolute Neutrophil Count (NEUTS) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Absolute Neutrophil Count (NEUTS)
Absolute Lymphocyte Count (LYMP) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Absolute Lymphocyte Count (LYMP)
Absolute Monocyte Count (MONO) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Absolute Monocyte Count (MONO)
Absolute Eosinophil Count (EOS) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Absolute Eosinophil Count (EOS)
Absolute Basophil Count (BASO) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Absolute Basophil Count (BASO)
Red Cell Distribution Width (RDW) | Measured at baseline and end-of-study (28 days)
  The effect of Actazin High Dose, Actazin Low Dose, Livaux High Dose, Livaux Low Dose, Control Formula, and placebo on Red Cell Distribution Width (RDW)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Clinical Trial Centers, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided